CLINICAL TRIAL: NCT01756352
Title: Assessment of the Utility of the Radiotracer "FET"in PET Imaging of Recurrent Glioblastoma Multiforme (GBM): Monitoring Early Response to Antiangiogenic Therapy
Brief Title: FET-PET for Evaluation of Response of Recurrent GBM to Avastin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marcelo F. Di Carli, MD, FACC (Other)
Responsible Party: Sponsor-Investigator, Marcelo F. Di Carli, MD, FACC, Chief of Nuclear Medicine/PET, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012P002678
Record Dates: First submitted 2012-12-20; First posted 2012-12-25 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Glioblastoma Multiforme; GBM
Keywords: FET; Fluoroethyl tyrosine; GBM; Response to treatment; Avastin; Brain Tumor
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — (18F)fluoroethyltyrosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GBM Avastin receiving 18F-FET (Experimental): Recurrent GBM patients receiving Avastin, imaged twice with 18F-FET PET before and approximately 8 weeks after receiving Avastin
  Interventions: Drug: 18F-FET

INTERVENTIONS:
Drug: 18F-FET — Radiotracer, surrogate marker for protein synthesis
  Other Names: 18F-Fluoroethyltyrosine

SUMMARY:
Hypothesis: The central hypothesis underlying the proposed research study is that FET-PET will predict durable benefit in patients receiving anti-angiogenic benefit for presumed recurrent GBM (i.e. progression-free survival and overall survival). We have defined one primary specific aim, for which we expect to obtain definitive results, and two secondary aims, under which we plan to generate preliminary data to support a future, larger project.

DETAILED DESCRIPTION:
The PET radiotracer FET provides a measure of large, neutral amino acid transport. This transport is significantly upregulated in malignant brain tumors. FET rarely gives false positive findings in the setting of inflammation seen after high dose chemotherapy or radiotherapy. FET labels low-grade as well as high-grade gliomas, in contrast to FDG, which almost exclusively labels only high-grade gliomas. FET imaging may prove to be particularly useful in the setting of infiltrative tumor, which is not contrast-enhancing on MRI and therefore not detectable with FDG. Management of glioblastoma patients with stable contrast-enhancing disease on MRI but increased signs of edema is difficult. This is because it is difficult to distinguish simple edema from infiltrative tumor. The former is managed with steroids and the latter is managed with chemotherapy, and anti-angiogenic drugs.

FET may be particularly useful in assessing changes after GBM patients receive anti-vascular agents such as Avastin. Avastin is very commonly used in patients after failure of first-line treatment in GBM. Not only is Avastin costly, but it also can have serious side effects such as internal bleeding and gastric perforation, severe hypertension, poor wound healing, and renal toxicity. It is important to know when a patient is failing Avastin treatment so that the drug can be discontinued. Preliminary data in Europe (see figures below) suggests that FET-PET can accurately distinguish Avastin responders from non-responders.

Inclusion Criteria:

1. GBM patients with changes on MRI suggestive of recurrence who have not yet initiated antiangiogenic therapy.
2. Age ≥ 18
3. Anticipated survival >3 months
4. Able to give informed consent
5. Capable of undergoing scan without the need for sedation or general anesthesia.

Exclusion Criteria:

1. Active intracranial infection or nonglial brain mass.
2. Recent large intracranial hemorrhage (<1 month; size to be determined by principal investigator)
3. Pregnant or nursing. Quantitative serum hCG testing will be performed prior to the initial and each -subsequent FET- PET scan on all females of childbearing potential. Our BWH Radiation Safety Committee and Partners IRB requires stat serum ß-hcG pregnancy tests.
4. Patient lives too far from BWH and/or is unwilling/ unable to return for scheduled imaging visits.

ELIGIBILITY:
Inclusion Criteria:

* 1. GBM patients with changes on MRI suggestive of recurrence who have not yet initiated antiangiogenic therapy. 2. Age ≥ 18 3. Anticipated survival >3 months 4. Able to give informed consent 5. Capable of undergoing scan without the need for sedation or general anesthesia.

Exclusion Criteria:

1. Active intracranial infection or nonglial brain mass.
2. Recent large intracranial hemorrhage (<1 month; size to be determined by principal investigator)
3. Pregnant or nursing. Quantitative serum hCG testing will be performed prior to the initial and each -subsequent FET- PET scan on all females of childbearing potential. Our BWH Radiation Safety Committee and Partners IRB requires stat serum ß-hcG pregnancy tests.
4. Patient lives too far from BWH and/or is unwilling/ unable to return for scheduled imaging visits.

   -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-02; Primary Completion 2015-09-13 (Actual); Study Completion 2015-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond L Huang, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GBM Avastin Receiving 18F-FET
Started | 13
Completed | 12
Not Completed | 1
Not completed — moved away and lost to followup | 1

BASELINE CHARACTERISTICS:
Arm/Group | GBM Avastin Receiving 18F-FET
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 61.4 [18 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: The primary objective is to assess the utility of FET-PET imaging for prediction of progression-free survival in recurrent glioblastoma.
Time Frame: From date of baseline PET scan until the date of death from any cause, assessed up to 2 years.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | GBM Avastin Receiving 18F-FET
Number analyzed (Participants) | 12
days | 158.25 (161.7)

2. Secondary Outcome: Overall Survival
Description: The secondary objective is to assess the utility of FET-PET imaging for prediction of overall survival in recurrent glioblastoma.
Time Frame: From date of baseline PET scan until the date of death from any cause, assessed up to 2 years.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | GBM Avastin Receiving 18F-FET
Number analyzed (Participants) | 12
days | 270.58 (222.00)

ADVERSE EVENTS:
Time Frame: From date of baseline PET scan until the date of death from any cause, assessed up to 2 years.
Arm/Group | GBM Avastin Receiving 18F-FET
All-Cause Mortality (participants affected / at risk) | 12/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GBM Avastin Receiving 18F-FET (N=12)
Bruising (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No